CLINICAL TRIAL: NCT02136277
Title: Measurement of Changes in Macro- and Microvascular Blood Flow During Major Colorectal Surgery
Brief Title: Vascular Changes During Colorectal Surgery
Acronym: MaMiFlo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Thomas Heinink, Clinical research fellow in anaesthesia, University of Nottingham
Other Study IDs: 13115
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Patients Undergoing Open Resection of Colorectal Tumours
Keywords: colorectal surgery; cardiac output
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal patients: Subjects undergoing colorectal surgery
  Interventions: Drug: Hartmann's solution

INTERVENTIONS:
Drug: Hartmann's solution — Administered in 250ml boluses, until cardiac output has been optimised.
  Other Names: Compound sodium lactate solution; Ringer's lactate solution; Lactated Ringer's solution

SUMMARY:
The purpose of this study is to investigate whether increases in the blood flow from the heart (the cardiac output), induced by the administration of intravenous fluids, lead to an increase in the blood flow to the vital organs, in patients undergoing bowel surgery.

This study will involve 2 phases. Firstly, potential volunteers will be invited to meet the research fellow (medical doctor) undertaking this study, who will check their suitability to participate in the study and who will obtain informed consent.

The second phase is the study itself which will take place whilst volunteers are having their bowel operation. They will attend theatre in the normal way, but once they have been anaesthetised (put to sleep), a special monitor called an oesophageal doppler probe will be placed into their oesophagus (food pipe) via the nose. This monitor is frequently used in bowel surgery to help assess how much intravenous fluid to administer to a patient by measuring the cardiac output (the amount of blood pumped out of the heart each minute). Using the cannula (drip) already inserted in the arm to allow administration of the anaesthetic, a special fluid, called an ultrasound contrast agent, will be injected into the drip, to allow a contrast enhanced ultrasound scan of the abdominal organs to be performed, to measure the blood flow to these organs. A small sample of blood will be taken from the earlobe to allow us to measure a chemical in the blood called lactate.

After this, intravenous fluid will be administered in order to increase the amount of blood pumped out of the heart. Once the oesophageal doppler monitor suggests that an adequate amount of fluid has been given, a second ultrasound scan will be performed to measure whether blood flow to the abdominal organs has also increased. A further blood sample will be taken from your earlobe to measure any change in lactate level.

At the completion of the operation, a third ultrasound scan will be performed and another sample of blood taken from the earlobe, to help assess blood flow to the organs.

DETAILED DESCRIPTION:
Potential participants (patients with colorectal cancer offered an operation) will be highlighted from the Derbyshire NHS trusts colorectal multidisciplinary team meeting. All patients who fulfil entry requirements will be seen by the research fellow after their outpatient meeting with their particular surgeon (if they agree). Information packs containing details of the study (information sheet and consent form) will be given and any questions answered. Patients will be allowed to take the packs away with them and decide whether they would be keen to participate. Interested patients will be consented by the research fellow during their subsequent pre-operative clinic appointment.

The study will take place intra-operatively. Monitoring will be instituted as determined necessary by the attending anaesthetists, but as a minimum will consist of pulse oximetry, ECG and non-invasive blood pressure recording. Intravenous cannulae will be sited and general anaesthesia induced by the anaesthetist responsible for the patient, as would be normal for this type of surgery. Once the patient has been transferred to the operating theatre, the research fellow will insert an ODM probe via either the nasal or oral route and the CO and SV will be measured; this constitutes normal care. A sterile Phillips iU22 USS probe will be placed on the patient's abdomen and the research fellow will administer SonoVue contrast agent intravenously via the cannula already sited to facilitate anaesthesia, up to a maximum dose of 2.4ml. Visceral MVBF will be measured using this CEUS technique. Capillary blood samples will be taken from earlobe for measurement of blood lactate levels by the research fellow. At this stage, as would typically occur during an operation of this nature, the research fellow will administer intravenous colloid suspension in boluses of 3ml/kg, up to a maximum of 15ml/kg, until the CO has been maximised, as judged by the ODM. At this stage, the research fellow will perform a further CEUS of the abdominal viscera by administering Sonovue contrast agent (2nd dose of up to 2.4ml) and measuring MVBF with the Phillips iU22. Repeat samples of capillary blood will be drawn to measure the lactate level by the research fellow. At the end of the operation, a 3rd CEUS of the abdominal viscera, along with further SV & CO readings, will be made.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 80 years
* Confirmed colorectal cancer
* Offered surgery by Derbyshire colorectal multidisciplinary team
* No metastatic disease
* Able to consent in English by themselves

Exclusion Criteria:

* Metastatic disease
* Oesophageal varices
* Patients with recent acute coronary syndrome (symptoms involving the heart) or unstable ischaemic cardiac disease (reduced blood supply to the heart);
* Patients known to have right-to-left shunts (abnormal movement of blood within the heart), severe pulmonary hypertension (high blood pressure in the pulmonary artery, the blood vessel that leads from the heart to the lungs), uncontrolled hypertension (high blood pressure) or adult respiratory distress syndrome (severe fluid build-up in both lungs);
* Pregnant or breast-feeding women;
* Known sensitivity to Sonovue;
* Prolonged QT syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancers, scheduled to undergo open resectional surgery.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Changes in microvascular blood flow during colorectal surgery | Immediately following optimisation of cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: John P Williams, PhD, Study Chair — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom